CLINICAL TRIAL: NCT02762617
Title: Phase 1 Safety and Pharmacokinetic Study of a Polyurethane Tenofovir Disoproxil Fumarate Vaginal Ring in Sexually Active Women (TDF IVR-002)
Brief Title: Safety and Pharmacokinetics (PK) of a Polyurethane Tenofovir Disoproxil Fumarate (TDF) Vaginal Ring (TDF IVR-002)
Acronym: TDF IVR-002
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety-related
Sponsor: Marla Keller (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Marla Keller, Professor, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-5591; U19AI103461 (NIH)
Record Dates: First submitted 2016-04-22; First posted 2016-05-05 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy; HIV
Keywords: Healthy Volunteers; Women's Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TDF IVR group (Experimental): The Tenofovir Disoproxil Fumarate intravaginal ring (TDF-IVR) is a white (with clear segment), flexible torus-shaped device with an inner core which contains the experimental drug, TDF, and sodium chloride. The intravaginal ring is worn continuously for 28 days and replaced with new rings twice (every 28 days) for total of 84 days (3 months).
  Participants will be stratified by site and will be randomized in a 3:1 ratio (TDF:Placebo).
  Interventions: Drug: Tenofovir disoproxil fumarate intravaginal ring
- Placebo IVR group (Placebo Comparator): The placebo intravaginal ring (IVR) is a clear, flexible torus-shaped device with an inner core which contains sodium chloride. The intravaginal ring is worn continuously for 28 days and replaced with new rings twice (every 28 days) for total of 84 days (3 months).
  Participants will be stratified by site and will be randomized in a 3:1 ratio (TDF:Placebo).
  Interventions: Drug: Placebo intravaginal ring (IVR)

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate intravaginal ring — The TDF IVR is formulated using preformed flexible tubing, comprised of biomedical medical grade hydrophilic, aliphatic polyurethane, and an inner core compartment comprised of 86% (w/w) TDF and 14% (w/w) sodium chloride. The ring will be inserted by the study clinician and worn for 28 day intervals for a total of 3 months (84 days). The ring will be removed and replaced with a new ring at each 28 day interval.
  Other Names: TDF IVR
  Arms: TDF IVR group
Drug: Placebo intravaginal ring (IVR) — The Placebo IVR is formulated using preformed flexible tubing, comprised of biomedical medical grade hydrophilic, aliphatic polyurethane, and an inner core compartment comprised of sodium chloride. The ring will be inserted by the study clinician and worn for 28 day intervals for a total of 3 months (84 days). The ring will be removed and replaced with a new ring at each 28 day interval.
  Other Names: Placebo
  Arms: Placebo IVR group

SUMMARY:
This prospective, two-site, two-arm, randomized, single-blind, placebo-controlled trial will examine the safety and pharmacokinetics (PK) of a polyurethane tenofovir disoproxil fumarate (TDF) vaginal ring when used continuously for 84 consecutive days by sexually active women.

The primary objective is to assess the safety of TDF vaginal rings when used continuously for 84 days by healthy, HIV-uninfected, sexually active women, as compared with a placebo vaginal ring.

DETAILED DESCRIPTION:
Tenofovir disoproxil fumarate (TDF) is a prodrug of TFV, an adenosine nucleoside monophosphonate (nucleotide) derivative with potent antiretroviral (ARV) activity. TDF is licensed for the treatment of HIV-1 infection in the US, the European Union, Middle East, and Africa. TDF permeates cells more rapidly than TFV resulting in increased intracellular accumulation of TFV- diphosphate (TFV-DP), the active metabolite. TDF is more potent than TFV and inhibits HIV-1 and herpes simplex virus type 2 (HSV-2) infection in cell and tissue culture models at approximately 100-fold lower concentrations than TFV, suggesting that it may be an excellent candidate for prevention of HIV.

The study will take place at the Albert Einstein College of Medicine in Bronx, USA and the Thick Partners Study Clinic (Partners in Health Research and Development) in Thika, Kenya. This is the the second clinical study of the polyurethane TDF vaginal ring (TDF IVR-002) following the successful completion of a first-in-human study (TDF IVR-001). It is hypothesized that the TDF IVR will be safe and well tolerated among healthy, sexually active women in the US and Kenya. It is also hypothesized that there will be a favorable PK profile in sexually active women. The null hypothesis is that there will be no difference in the safety profile between the active product and the placebo.

Each participant will receive an IVR containing TDF or a placebo ring. The vaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses, by the study clinician at Visit 3 and removed by the study clinician at Visit 7. Each participant will be followed for 7 days following ring removal.

Building on the results of the first TDF IVR study in sexually abstinent women, a longer Phase 1 study was designed in order to assess the safety and PK of TDF IVR in sexually active women. Vaginal rings have been tested in several clinical trials in women 18 years of age and older and have been found to be safe. Given the drug release kinetics observed in vitro, in preclinical studies, and in the first Phase 1 study, TDF and TFV (formed following hydrolysis of the prodrug TDF) concentrations in CVF are expected to reach steady state within one day and within one month for tissue and maintain steady state concentrations for the duration of the planned 84 days of ring use. Sampling at multiple time points will provide information on drug kinetics, and, by sampling after ring removal how long drug persists. The latter may be important as behavior studies suggest that some women may remove a ring at time of menses or around sex. Tissue sampling in US women in the hours and days immediately following ring insertion will provide valuable information about early tissue levels and the time required to achieve drug concentrations needed for protection. To capture systemic absorption, blood will be sampled to determine drug concentrations in plasma and DBS. To capture the concentrations of drug within the genital tract, CVF will be collected from the posterior fornix using Dacron swabs. Cervical tissue sampling will be highly informative given that it is the likely site of drug action. However, biopsies must be taken sparingly as they are uncomfortable to some and alter the healing process. Accordingly, 2 biopsies for PK studies will be obtained in US women at Days 28 and 56 when the ring is changed, and at Day 84 when the final ring is removed. US women will also have an additional 2 biopsies collected at only 1 of 7 time-points (5 or 6 women per time-point at either 1 hour, 4 hours, 1, 7, 14, or 21 days after ring insertion, or 5-7 days after ring removal). Participants in Kenya will have 2 cervical biopsies collected at each of 2 study visits (Days 28 and 84). The study will be single-blinded because the TDF and placebo rings are not identical in appearance. All participants will be informed that 2 biopsies will be taken during study visits in which biopsies will be collected. Cervical biopsies will be obtained without local anesthetic. Participants may take acetaminophen before and/or after the biopsies are collected, if desired. Participants will be instructed to abstain from sex for 7 days after biopsy collection to allow adequate time to heal.

Primary Objective:

• Assess the safety of TDF IVR when used continuously for 84 days by healthy, HIV-uninfected, sexually active women, as compared with the placebo IVR

Secondary Objectives:

* Examine systemic and genital tract PK of TDF release during and after 84 days of continuous IVR use in sexually active women
* Evaluate the acceptability of the study IVR in HIV-uninfected, sexually active women over 84 days of use

This is a two-site, two-arm, randomized single blind placebo-controlled trial. The study population will include approximately 80 healthy, 18-45 year old females who are HIV-uninfected, non-pregnant, non-breastfeeding, sexually active and using contraception. Forty US women and 40 Kenyan women will be stratified by site and will be randomized 3:1 (30 TDF:10 placebo at each site).

The Kenya site will not initiate enrollment until an interim analysis is performed on the first 20 US women who have completed 30 days of ring use. Enrollment at both sites will include women using a copper intrauterine device (IUD) or a hormonal contraceptive method other than an IVR. To ensure participants are protected from pregnancy and sexually transmitted infections (STI) during study participation, condoms will be distributed at each study visit. As this is a Phase 1 trial of a TDF IVR, only healthy women with a low risk profile for HIV will be recruited and will be asked to wear a TDF or placebo IVR for 84 days. Participants will be strongly encouraged to include their male partner in the study. If participants are willing, education and counseling will be provided to male partners at all study visits and up to 20 males at the Thika site will be invited to participate in qualitative interviews if able and willing to provide written informed consent.

The approximate time to complete study enrollment is expected to be 12 months. Given the need to carefully screen and exclude women who are not able to comply to study procedures, we anticipate that the Thika site will not enroll more than 1 participant per week. Two study groups are planned at each site. All groups will be assigned to complete a total of 9 study visits (Screening [visit 1], Enrollment [visit 2], Day 14 [visit 3], 28 [visit 4], 42 [visit 5], 56 [visit 6], 70 [visit 7], 84 [visit 8], 89 [visit 9]). Each US participant will be asked to undergo additional PK sampling at one of the following time-points: either 1 hour (visit 2a), 4 hours (visit 2b), 1 (visit 2c), 7 (visit 2d), 14 (visit 3a), or 21 days (visit 3b) after ring insertion, or 5-7 (visit 9a) and 10-12 days (visit 10) after ring removal.

The two study groups are:

1. Reservoir-type polyurethane TDF IVR group;
2. Reservoir-type polyurethane Placebo IVR group;

The expected duration for participants is approximately 120 days (including a screening visit, an enrollment visit, 84 days of continuous IVR use, and 5-7 days following IVR removal). Participants will undergo Visit 2 within 28 days of screening. No study data will be collected after the Final Study/Early Termination Visit unless the participant is pregnant at the Final Study/Early Termination Visit. Participants who have AEs at the Final Study/Early Termination Visit that have not resolved or stabilized will be followed beyond the Final Study/Early Termination Visit until a clinically acceptable resolution of the AE(s) is confirmed and documented. Clinical acceptability of resolution will be determined by the Project Leader (PL) in consultation with the Protocol Safety Review Team (PSRT). Participants identified as infected with HIV during the study will be managed in accordance with the study protocol. Participants who are pregnant at the Final Study/Early Termination Visit may be followed in accordance with procedures described in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years (inclusive) at screening.
* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes).
* Able and willing to provide written informed consent to be screened for and take part in the study.
* Able and willing to provide adequate locator information.
* Able and willing to avoid receptive vaginal and anal intercourse for 1 week after each biopsy.
* HIV-uninfected based on testing performed by study staff during screening procedures (per applicable algorithm in Appendix II).
* Using a copper IUD or any hormonal contraceptive method, other than an IVR, for a minimum of 2 months and intending to use the same method for the duration of study participation.
* Per participant report, sexually active, defined as having vaginal intercourse at least once in the month prior to screening.
* Have a regular sex partner and willing to have at least 4 sex acts per month for the duration of the study. Sex act is defined as penile-vaginal penetrative intercourse. Study staff will provide condoms to all study participants. Participants will not be restricted from engaging in oral sex.
* Has not used pre- or post-exposure prophylaxis for HIV exposure in the 3 months prior to Screening.
* Per participant report at Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products for the duration of study participation.
* At Screening, participant states she is able and willing to refrain from taking traditional herbs or medicines and is willing to refrain from inserting any non-study vaginal products or objects into the vagina, including but not limited to, spermicides, diaphragms, contraceptive vaginal rings, vaginal medications, vaginal probiotics/pre-biotics, menstrual cups, cervical caps (or any other vaginal barrier method), douches, lubricants, vaginal drying agents and sex toys (vibrators, dildos, etc.). Tampons may be used, but for menses only.
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection.

Exclusion Criteria:

Women must meet none of the following criteria prior to genital sampling at Enrollment:

Participant report of any of the following at Screening:

* Sex in the past 3 months or any possibility of sex during study participation with a partner who is HIV+ or with a partner of unknown HIV status.
* Known adverse reaction to polyurethane or to any components of the study product or allergy to both silver nitrate and Monsel's solution.
* Active hepatitis B infection.
* Chronic, recurrent, and/or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.).
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy.
* Intending to become pregnant during the period of study participation.
* Currently breastfeeding or planning to breastfeed during the course of the study.
* Menopause.
* History of unexplained or unresolved intermenstrual bleeding in the 3 months prior to screening.
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix in the last 14 days.
* Hysterectomy.
* Women using contraceptive IVRs because the study product is an IVR.
* Systemic use in the last 2 weeks or anticipated use during the study period of any of the following: corticosteroids, anticoagulants or ARVs.
* Plans to relocate away from the study site area during the period of study participation.
* Grade 1 or higher laboratory abnormality, as defined by the DAIDS Table for Grading the Severity of Adult and Pediatric AEs, Version 2.0, Nov 2014.
* At Screening or Enrollment, is pregnant (based on urine pregnancy test).
* In the last three months, diagnosed with or treated for any STI. Note: Women with a history of condylomata or genital herpes may be considered for eligibility as long as there are no lesions on exam. HSV 1 and 2 serologies will be obtained. Participants will be included regardless of the results of these serologies.
* Reproductive tract infection (RTI) or pelvic inflammatory disease (PID) requiring treatment per local guidelines in Kenya and Centers for Disease Control and Prevention (CDC) guidelines in the US at Screening or Enrollment.

Note: Otherwise eligible women diagnosed with symptomatic vulvovaginal candidiasis (VVC), symptomatic bacterial vaginosis (BV) or urinary tract infection (UTI) will be eligible if Visit 2 (Enrollment) is scheduled after all symptoms have resolved and at least two weeks after completing treatment. Women with recurrent VVC and symptomatic BV despite treatment will be offered another course of treatment and will not be eligible.

* Positive test for Trichomonas vaginalis, Neisseria gonorrhea or Chlamydia trachomatis at screening.
* Positive test for hepatitis B (defined as positive for hepatitis B surface antigen).
* Reactive serologic test for syphilis at screening (per local guidelines). Note: Women with a history of syphilis that was not acquired and/or treated within the past 3 months and that has been appropriately treated may be considered for eligibility.
* At Screening or Enrollment, has a clinically apparent Grade 1 or higher pelvic exam finding (observed by study clinician or designee) per the DAIDS Table for Grading the Severity of Adult and Pediatric AEs, Addendum 1, Female Genital Grading Table for Use in Microbicide Studies.

Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the PL/designee is considered expected non-menstrual bleeding and is not exclusionary.

- Pap result Grade 2 or higher according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric AEs, Version 1.0, December 2004 (Clarification dated August 2009).

Note: Women 21 years of age or older with a documented normal result within the 12 months prior to enrollment need not have Pap smear during the screening period. Women with a Grade 1 abnormal Pap smear can be enrolled upon completion of the initial phase of evaluation if no current treatment is indicated (based on local standard of care for management of abnormal cervical cytology). Need for a repeat Pap within 6 months does not preclude enrollment prior to that result becoming available.

* At Screening, has severe pelvic relaxation such that either the vaginal walls or the uterine cervix descend beyond the vaginal introitus with Valsalva maneuver.
* Has any condition that, in the investigator's opinion, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Proportion of women in each arm experiencing adverse events (AEs) | Duration of study - 12 weeks (84 days)
  Genitourinary events Grade 2 or higher as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events judged to be related to study product.
  Adverse events Grade 2 or higher as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

SECONDARY OUTCOMES:
Assessment of TDF levels in cervicovaginal fluid (CVF) - Cmax | Days 28, 42, 56, 70, and 84 after TDF ring insertion
  Analysis for routine PK parameters: Maximum Concentration (Cmax)
Assessment of TDF levels in cervicovaginal fluid (CVF) - Tmax | Days 28, 42, 56, 70, and 84 after TDF ring insertion
  Analysis for routine PK parameters: Time to Maximum Concentration (Tmax)
Assessment of TDF levels in cervicovaginal fluid (CVF) - AUC | Days 28, 42, 56, 70, and 84 after TDF ring insertion
  Analysis for routine PK parameters: Area Under the Curve (AUC)
Assessment of TFV (tenofovir) levels in cervicovaginal fluid and plasma - Cmax | Days 28, 42, 56, 70, and 84 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV (tenofovir) levels in cervicovaginal fluid and plasma - Tmax | Days 28, 42, 56, 70, and 84 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV (tenofovir) levels in cervicovaginal fluid and plasma - AUC | Days 28, 42, 56, 70, and 84 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV-DP (tenofovir diphosphate) levels in dried blood spots (DBS) - Cmax | Days 28, 56, and 84 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV-DP (tenofovir diphosphate) levels in dried blood spots (DBS) - Tmax | Days 28, 56, and 84 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV-DP (tenofovir diphosphate) levels in dried blood spots (DBS) - AUC | Days 28, 56, and 84 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV levels in cervical tissue - Cmax | Days 28, 56 (US participants only), and 84 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV levels in cervical tissue - Tmax | Days 28, 56 (US participants only), and 84 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV levels in cervical tissue - AUC | Days 28, 56 (US participants only), and 84 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV-DP levels in cervical tissue - Cmax | Days 28, 56 (US participants only), and 84 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV-DP levels in cervical tissue - Tmax | Days 28, 56 (US participants only), and 84 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV-DP levels in cervical tissue - AUC | Days 28, 56 (US participants only), and 84 after TDF ring insertion
  Analysis for routine PK parameters (AUC)

OTHER OUTCOMES:
Assessment of TDF levels in CVF - Cmax | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TDF levels in CVF - Tmax | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TDF levels in CVF - AUC | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV levels in CVF and tissue - Cmax | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV levels in CVF and tissue - Tmax | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV levels in CVF and tissue - AUC | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV-DP levels in tissue - Cmax | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV-DP levels in tissue - Tmax | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV-DP levels in tissue - AUC | 1 Hour, 4 Hours, and Day 1 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV levels in plasma, CVF, and tissue - Cmax | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV levels in plasma, CVF, and tissue - Tmax | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV levels in plasma, CVF, and tissue - AUC | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TDF levels in CVF - Cmax | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TDF levels in CVF - Tmax | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TDF levels in CVF - AUC | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV-DP levels in tissue - Cmax | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (Cmax)
Assessment of TFV-DP levels in tissue - Tmax | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (Tmax)
Assessment of TFV-DP levels in tissue - AUC | Days 7, 14, and 21 after TDF ring insertion
  Analysis for routine PK parameters (AUC)
Assessment of TFV-DP levels in tissue - Cmax | 5-7 days after ring removal
  Analysis for routine PK parameters (Cmax)
Assessment of TFV-DP levels in tissue - Tmax | 5-7 days after ring removal
  Analysis for routine PK parameters (Tmax)
Assessment of TFV-DP levels in tissue - AUC | 5-7 days after ring removal
  Analysis for routine PK parameters (AUC)
Assessment of TDF levels in CVF - Cmax | 10-12 days after ring removal (US participants only)
  Analysis for routine PK parameters (Cmax)
Assessment of TDF levels in CVF - Tmax | 10-12 days after ring removal (US participants only)
  Analysis for routine PK parameters (Tmax)
Assessment of TDF levels in CVF - AUC | 10-12 days after ring removal (US participants only)
  Analysis for routine PK parameters (AUC)
Assessment of TFV levels in CVF and plasma - Cmax | 10-12 days after ring removal (US participants only)
  Analysis for routine PK parameters (Cmax)
Assessment of TFV levels in CVF and plasma - Tmax | 10-12 days after ring removal (US participants only)
  Analysis for routine PK parameters (Tmax)
Assessment of TFV levels in CVF and plasma - AUC | 10-12 days after ring removal (US participants only)
  Analysis for routine PK parameters (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Marla J Keller, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- Albert Einstein College of Medicine, The Bronx, New York, United States
- Kenya Medical Research Institute, Partners in Prevention, University of Nairobi, Nairobi, Kenya

REFERENCES:
- [Result] Keller MJ, Mesquita PM, Marzinke MA, Teller R, Espinoza L, Atrio JM, Lo Y, Frank B, Srinivasan S, Fredricks DN, Rabe L, Anderson PL, Hendrix CW, Kiser PF, Herold BC. A phase 1 randomized placebo-controlled safety and pharmacokinetic trial of a tenofovir disoproxil fumarate vaginal ring. AIDS. 2016 Mar 13;30(5):743-51. doi: 10.1097/QAD.0000000000000979. PMID 26605514
- [Derived] Keller MJ, Wood L, Billingsley JM, Ray LL, Goymer J, Sinclair S, McGinn AP, Marzinke MA, Frank B, Srinivasan S, Liu C, Atrio JM, Espinoza L, Mugo N, Spiegel HML, Anderson PL, Fredricks DN, Hendrix CW, Marrazzo J, Bosinger SE, Herold BC. Tenofovir disoproxil fumarate intravaginal ring for HIV pre-exposure prophylaxis in sexually active women: a phase 1, single-blind, randomised, controlled trial. Lancet HIV. 2019 Aug;6(8):e498-e508. doi: 10.1016/S2352-3018(19)30145-6. Epub 2019 Jul 15. PMID 31320290